CLINICAL TRIAL: NCT02583256
Title: A Phase III, Randomized, Observer Blind, Multicenter Study to Evaluate the Safety and Immunogenicity of Repeated Exposure to Either the Same or Alternate Type of Vaccine, Adjuvanted or Non-adjuvanted Quadrivalent Subunit Influenza Virus Vaccine (aQIV or QIV), Administered to Subjects Previously Vaccinated in Trial V118_05 (NCT01964989)
Brief Title: Clinical Study to Evaluate Safety, Immunogenicity of Investigational Flu Vaccine Compared to an Approved Flu Vaccine in Children Previously Vaccinated in Trial V118_05 (NCT01964989)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V118_05E3; 2015-002973-39 (EudraCT Number)
Record Dates: First submitted 2015-10-16; First posted 2015-10-22 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Influenza
Keywords: Influenza Vaccine; MF59 adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- aQIV/aQIV (Experimental): Subjects previously vaccinated with aQIV followed one year later by aQIV
  Interventions: Biological: Adjuvanted QIV (aQIV)
- aQIV/QIV (Experimental): Subjects previously vaccinated with aQIV followed one year later by QIV
  Interventions: Biological: Non-adjuvanted QIV
- QIV/aQIV (Experimental): Subjects previously vaccinated with QIV followed one year later by aQIV
  Interventions: Biological: Adjuvanted QIV (aQIV)
- QIV/QIV (Experimental): Subjects previously vaccinated with QIV followed one year later by QIV
  Interventions: Biological: Non-adjuvanted QIV

INTERVENTIONS:
Biological: Adjuvanted QIV (aQIV) — Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine (aQIV)
  Arms: QIV/aQIV; aQIV/aQIV
Biological: Non-adjuvanted QIV — Non-adjuvanted Quadrivalent Influenza Vaccine (QIV)
  Arms: QIV/QIV; aQIV/QIV

SUMMARY:
Safety, Immunogenicity of an Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine Compared to Non-Adjuvanted Comparator Influenza Vaccine in Children Previously vaccinated in Trial V118_05. Subjects will receive either the Same or Alternate Type of Vaccine.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, all subjects must meet ALL of the inclusion criteria described.

* Subject's parent/legal guardian has voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
* Male or female subject who has completed their Visit 13 (Study Day 366 for non-naïve subjects) or clinic Visit 15 (Day 390 for naïve subjects) in parent trial V118_05.
* For naïve subjects in parent trial V118_05 to have received two doses of the same study vaccine (i.e. 2 doses of aQIV or 2 doses of QIV).

Exclusion Criteria:

* Previous immunization with any influenza vaccine (licensed or investigational) within 6 months prior to enrollment.
* Subjects with a clinical condition representing a contraindication to intramuscular vaccination or blood draws.
* Unwillingness of the parent(s)/ legal guardian(s) of the subject to refuse to participate in another clinical trial while enrolled in V118-05E3.

Additional eligibility criteria may be discussed by contacting the site.

Ages: 12 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1601 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (17):
- Finland (9):
  - Investigational Site- 001, Espoo, Etelä-Suomen Lääni
  - Investigational Site- 002, Helsinki, Etelä-Suomen Lääni
  - Investigational Site- 003, Helsinki, Etelä-Suomen Lääni
  - Investigational Site- 004, Jarvenpaa, Etelä-Suomen Lääni
  - Investigational Site- 005, Kokkola, Länsi-Suomen Lääni
  - Investigational Site- 007, Pori, Länsi-Suomen Lääni
  - Investigational Site- 009, Tampere, Länsi-Suomen Lääni
  - Investigational Site- 010, Turku, Länsi-Suomen Lääni
  - Investigational Site- 006, Oulu
- Philippines (4):
  - Investigational Site- 303, Laguna, Matro Manila
  - Investigational Site- 304, Muntinlupa, National Capital Region
  - Investigational Site- 305, Muntinlupa, National Capital Region
  - Investigational Site- 306, Cavite
- Thailand (4):
  - Investigational Site- 325, Pathum Thani, Bangkok
  - Investigational Site- 320, Bangkok, Changwat Samut Prakan
  - Investigational Site- 327, Bangkok, Krung Thep Maha Nakhon [Bangko
  - Investigational Site- 323, Bangkok

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 17 sites in total; 9 sites in Finland, 4 sites in the Philippines and 4 sites in Thailand.
Pre-assignment Details: All enrolled subjects were included in the study.
Period: Overall Study
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Started | 403 | 403 | 402 | 393
Exposed | 403 | 403 | 402 | 393
Completed | 400 | 401 | 400 | 390
Not Completed | 3 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — Administrative/Other | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV | Total
Number analyzed (Participants) | 403 | 403 | 402 | 393 | 1601
Age, Continuous [Mean (Standard Deviation); unit: months] | 54.4 (17.12) | 52.3 (17.02) | 53.4 (17.32) | 53.3 (17.30) | 53.0 (16.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 189 | 206 | 178 | 770
  Male | 206 | 214 | 196 | 215 | 831
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 402 | 403 | 402 | 392 | 1599
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 364 | 364 | 362 | 355 | 1445
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 38 | 36 | 37 | 35 | 146
  Other | 1 | 3 | 3 | 3 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Philippines | 210 | 211 | 213 | 212 | 846
  Finland | 39 | 39 | 39 | 38 | 155
  Thailand | 154 | 153 | 150 | 143 | 600
Risk Status [Count of Participants; unit: Participants] — Subjects with underlying conditions that posed high risk of influenza complications (at risk/not at risk)
  Participants
    At risk | 10 | 20 | 18 | 13 | 61
    Not at risk | 393 | 383 | 384 | 380 | 1540

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) and GMT Ratio as Determined by Hemagglutination Inhibition (HI) Assay on Day 22 Against Homologous Strains (aQIV-primed Comparison), Noninferiority Analysis
Description: GMT and 95% confidence interval (CI) were analyzed for Day 22 against homologous strains using ANCOVA with study specific covariates.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 22
Population: Immunogenicity per protocol set (PPS) consisting of all subjects who received a study vaccination and provided immunogenicity data, and who correctly received the study vaccine, had no major protocol deviations, and did not develop reverse transcription polymerase chain reaction(RT-PCR) confirmed influenza infection between baseline and Visit 2.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | aQIV/aQIV | aQIV/QIV
Number analyzed (Participants) | 403 | 398
titer
  A/H1N1 | 1219.00 [1137.35 to 1306.52] | 1020.89 [953.22 to 1093.36]
  A/H3N2 | 2355.52 [2226.19 to 2492.35] | 2529.83 [2392.90 to 2674.59]
  B/Yamagata | 276.23 [252.73 to 301.92] | 232.82 [213.25 to 254.19]
  B/Victoria | 388.35 [355.33 to 424.44] | 328.42 [300.76 to 358.63]
Statistical Analysis 1: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain A/H1N1; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.19, 95% CI 2-sided [1.1 to 1.3]
Statistical Analysis 2: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain A/H3N2; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should not fall below 0.667; GMT ratio = 0.93, 95% CI 2-sided [0.9 to 1.0]
Statistical Analysis 3: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain B/Yamagata; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.19, 95% CI 2-sided [1.1 to 1.3]
Statistical Analysis 4: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain B/Victoria; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.18, 95% CI 2-sided [1.1 to 1.3]

2. Primary Outcome: Immunogenicity Endpoint: GMT and GMT Ratio as Determined by HI Assay on Day 22 Against Homologous Strains (aQIV-primed Comparison), Superiority Analysis
Description: GMT and 95% CI were analyzed for Day 22 against homologous strains using ANCOVA with study specific covariates.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 22
Population: The immunogenicity full analysis set (FAS) consisting of all subjects who received a study vaccination and provided immunogenicity data at both Visit 1 (baseline) and at least one post-vaccination visit.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | aQIV/aQIV | aQIV/QIV
Number analyzed (Participants) | 403 | 403
titer
  A/H1N1 | 1218.91 [1137.02 to 1306.70] | 1023.37 [955.72 to 1095.81]
  A/H3N2 | 2345.71 [2216.84 to 2482.07] | 2521.60 [2385.43 to 2665.56]
  B/Yamagata | 274.75 [251.09 to 300.65] | 230.51 [210.97 to 251.86]
  B/Victoria | 387.35 [354.15 to 423.66] | 326.68 [299.10 to 356.81]
Statistical Analysis 1: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain A/H1N1; Test type: Superiority — Superiority criterion for the GMT ratio: Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should exceed 1; GMT ratio = 1.19, 95% CI 2-sided [1.1 to 1.3]
Statistical Analysis 2: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain A/H3N2; Test type: Superiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should exceed 1; GMT ratio = 0.93, 95% CI 2-sided [0.9 to 1.0]
Statistical Analysis 3: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain B/Yamagata; Test type: Superiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should exceed 1; GMT ratio = 1.19, 95% CI 2-sided [1.1 to 1.3]
Statistical Analysis 4: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain B/Victoria; Test type: Superiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should exceed 1; GMT ratio = 1.19, 95% CI 2-sided [1.1 to 1.3]

3. Secondary Outcome: Immunogenicity Endpoint: GMT and GMT Ratio as Determined by HI Assay on Day 22 Against Homologous Strains (QIV-primed Comparison)
Description: as for outcome 2
Time Frame: Day 22
Population: The immunogenicity PPS consisting of all subjects who received a study vaccination and provided immunogenicity data, and who correctly received the study vaccine, had no major protocol deviations, and did not develop RT-PCR-confirmed influenza infection between baseline and Visit 2.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 397 | 389
titer
  A/H1N1 | 1206.20 [1123.80 to 1294.65] | 866.51 [807.30 to 930.06]
  A/H3N2 | 2369.95 [2236.39 to 2511.48] | 2229.48 [2103.42 to 2363.10]
  B/Yamagata | 221.54 [202.12 to 242.82] | 156.01 [142.32 to 171.02]
  B/Victoria | 330.94 [302.38 to 362.21] | 244.03 [222.84 to 267.24]
Statistical Analysis 1: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain A/H1N1; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of QIV-aQIV/QIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.39, 95% CI 2-sided [1.28 to 1.51]
Statistical Analysis 2: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain A/H3N2; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of QIV-aQIV/QIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.06, 95% CI 2-sided [0.99 to 1.14]
Statistical Analysis 3: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain B/Yamagata; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of QIV-aQIV/QIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.42, 95% CI 2-sided [1.27 to 1.58]
Statistical Analysis 4: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain B/Victoria; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of QIV-aQIV/QIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.36, 95% CI 2-sided [1.22 to 1.51]

4. Secondary Outcome: Immunogenicity Endpoint: GMT and GMT Ratio as Determined by HI Assay on Day 181 Against Homologous Strains (aQIV-primed and QIV-primed Comparison)
Description: GMT and 95% CI were analyzed for Day 181 against homologous strains using ANCOVA with study specific covariates.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 181
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 398 | 397 | 389
titer
  A/H1N1 | 489.45 [449.93 to 532.45] | 411.72 [378.83 to 447.46] | 429.06 [393.73 to 467.57] | 307.36 [282.02 to 334.98]
  A/H3N2 | 1423.38 [1310.04 to 1546.52] | 1438.40 [1325.53 to 1560.89] | 1233.84 [1133.08 to 1343.56] | 1222.21 [1121.92 to 1331.46]
  B/Yamagata | 97.01 [88.67 to 106.13] | 86.43 [79.09 to 94.45] | 73.37 [66.88 to 80.49] | 56.57 [51.56 to 62.08]
  B/Victoria | 128.32 [115.17 to 142.97] | 115.26 [103.57 to 128.26] | 104.93 [94.02 to 117.10] | 79.76 [71.41 to 89.09]
Statistical Analysis 1: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain A/H1N1; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.19, 95% CI 2-sided [1.07 to 1.32]
Statistical Analysis 2: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain A/H3N2; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should not fall below 0.667; GMT ratio = 0.99, 95% CI 2-sided [0.90 to 1.09]
Statistical Analysis 3: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain B/Yamagata; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.12, 95% CI 2-sided [1.01 to 1.25]
Statistical Analysis 4: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain B/Victoria; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of aQIV-aQIV/aQIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.11, 95% CI 2-sided [0.98 to 1.27]
Statistical Analysis 5: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain A/H1N1; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of QIV-aQIV/QIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.4, 95% CI 2-sided [1.3 to 1.5]
Statistical Analysis 6: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain A/H3N2; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of QIV-aQIV/QIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.01, 95% CI 2-sided [0.9 to 1.1]
Statistical Analysis 7: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain B/Yamagata; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of QIV-aQIV/QIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.30, 95% CI 2-sided [1.2 to 1.4]
Statistical Analysis 8: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain B/Victoria; Test type: Non-Inferiority — Lower bound of two-sided 95% CI on the ratio of QIV-aQIV/QIV-QIV HI GMT should not fall below 0.667; GMT ratio = 1.32, 95% CI 2-sided [1.2 to 1.5]

5. Secondary Outcome: Immunogenicity Endpoint: Seroconversion Rate (SCR) on Day 22 Against Homologous Strains (aQIV-primed and QIV-primed Comparison)
Description: The percentage of subjects achieving seroconversion at Day 22 after vaccination is reported against homologous strains. Seroconversion was defined in subjects seronegative at baseline (i.e. HI titer <1:10 on Day 1) as postvaccination HI titer ≥1:40 and defined in subjects seropositive at baseline (i.e. HI titer ≥1:10 on Day 1) as a minimum of a 4-fold increase in post-vaccination HI titer.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 1, Day 22
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 398 | 397 | 389
percentage of subjects
  A/H1N1 | 62.7 [57.8 to 67.4] | 60.9 [55.9 to 65.7] | 72.04 [67.35 to 76.40] | 62.37 [57.34 to 67.21]
  A/H3N2 | 68.9 [64.1 to 73.4] | 68.0 [63.2 to 72.6] | 72.80 [68.13 to 77.12] | 76.74 [72.21 to 80.86]
  B/Yamagata | 76.4 [71.9 to 80.4] | 72.0 [67.4 to 76.4] | 79.44 [75.11 to 83.32] | 66.49 [61.51 to 71.21]
  B/Victoria | 77.4 [73.0 to 81.4] | 74.8 [70.2 to 79.0] | 77.92 [73.49 to 81.92] | 69.55 [64.66 to 74.14]
Statistical Analysis 1: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain A/H1N1; Test type: Non-Inferiority — The lower bound of two-sided 95% CI on the difference between SCR should not be below -10%; SCR difference = 1.8, 95% CI 2-sided [-4.9 to 8.6]
Statistical Analysis 2: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain A/H3N2; Test type: Non-Inferiority — The lower bound of two-sided 95% CI on the difference between SCR should not be below -10%; SCR difference = 0.9, 95% CI 2-sided [-5.6 to 7.3]
Statistical Analysis 3: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain B/Yamagata; Test type: Non-Inferiority — The lower bound of two-sided 95% CI on the difference between SCR should not be below -10%; SCR difference = 4.3, 95% CI 2-sided [-1.8 to 10.4]
Statistical Analysis 4: Comparison: aQIV/aQIV vs aQIV/QIV; Comparison performed for strain B/Victoria; Test type: Non-Inferiority — The lower bound of two-sided 95% CI on the difference between SCR should not be below -10%; SCR difference = 2.6, 95% CI 2-sided [-3.3 to 8.5]
Statistical Analysis 5: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain A/H1N1; Test type: Non-Inferiority — The lower bound of two-sided 95% CI on the difference between SCR should not be below -10%; SCR difference = 9.67, 95% CI 2-sided [3.11 to 16.17]
Statistical Analysis 6: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain A/H3N2; Test type: Non-Inferiority — The lower bound of two-sided 95% CI on the difference between SCR should not be below -10%; SCR difference = -3.95, 95% CI 2-sided [-10.02 to 2.15]
Statistical Analysis 7: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain B/Yamagata; Test type: Non-Inferiority — The lower bound of two-sided 95% CI on the difference between SCR should not be below -10%; SCR difference = 12.95, 95% CI 2-sided [6.73 to 19.12]
Statistical Analysis 8: Comparison: QIV/aQIV vs QIV/QIV; Comparison performed for strain B/Victoria; Test type: Non-Inferiority — The lower bound of two-sided 95% CI on the difference between SCR should not be below -10%; SCR difference = 8.36, 95% CI 2-sided [2.17 to 14.54]

6. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) as Determined by HI Assay for Day 22/Day 1 and Day 181/Day 1 for Against Homologous Strains
Description: The GMR is the geometric mean of the fold increase in HI titer from Day 1 to Day 22 or Day 181. GMR and 95% CI were analyzed against homologous strains using ANCOVA with study specific covariates.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 22, Day 181
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 398 | 397 | 389
ratio
  A/H1N1 (Day 22/Day 1) | 7.69 [7.17 to 8.24] | 6.44 [6.01 to 6.90] | 7.61 [7.09 to 8.17] | 5.47 [5.09 to 5.87]
  A/H1N1 (Day 181/Day 1) | 3.11 [2.86 to 3.38] | 2.61 [2.40 to 2.84] | 2.72 [2.50 to 2.97] | 1.95 [1.79 to 2.13]
  A/H3N2 (Day 22/Day 1) | 9.02 [8.53 to 9.55] | 9.69 [9.17 to 10.25] | 9.08 [8.57 to 9.62] | 8.54 [8.06 to 9.05]
  A/H3N2 (Day 181/Day 1) | 5.44 [5.01 to 5.91] | 5.50 [5.07 to 5.97] | 4.72 [4.33 to 5.14] | 4.67 [4.29 to 5.09]
  B/Yamagata (Day 22/Day 1) | 7.81 [7.14 to 8.54] | 6.58 [6.03 to 7.19] | 6.26 [5.71 to 6.86] | 4.41 [4.02 to 4.83]
  B/Yamagata (Day 181/Day 1) | 2.74 [2.50 to 3.00] | 2.44 [2.23 to 2.67] | 2.07 [1.89 to 2.27] | 1.60 [1.46 to 1.75]
  B/Victoria (Day 22/Day 1) | 7.86 [7.19 to 8.59] | 6.64 [6.09 to 7.26] | 6.70 [6.12 to 7.33] | 4.94 [4.51 to 5.41]
  B/Victoria (Day 181/Day 1) | 2.59 [2.33 to 2.89] | 2.33 [2.09 to 2.59] | 2.12 [1.90 to 2.36] | 1.61 [1.44 to 1.80]

7. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects With HI Titer ≥1:40 on Day 22 and Day 181 Against Homologous Strains
Description: The percentage of subjects achieving HI titer ≥1:40 at Day 22 and Day 181 after vaccination is reported against homologous strains.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 22, Day 181
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 398 | 397 | 389
percentage of subjects
  A/H1N1 (Day 22) | 100 [99.1 to 100] | 100 [99.1 to 100] | 100 [99.1 to 100] | 99.7 [98.6 to 100]
  A/H1N1 (Day 181) | 100 [99.1 to 100] | 99.2 [97.8 to 99.8] | 99.2 [97.8 to 99.8] | 95.9 [93.4 to 97.6]
  A/H3N2 (Day 22) | 100 [99.1 to 100] | 100 [99.1 to 100] | 100 [99.1 to 100] | 100 [99.1 to 100]
  A/H3N2 (Day 181) | 99.8 [98.6 to 100] | 100 [99.1 to 100] | 100 [99.1 to 100] | 98.7 [97.0 to 99.6]
  B/Yamagata (Day 22) | 98.5 [96.8 to 99.5] | 98.7 [97.1 to 99.6] | 98.5 [96.7 to 99.4] | 96.6 [94.3 to 98.2]
  B/Yamagata (Day 181) | 94.3 [91.5 to 96.3] | 93.9 [91.1 to 96.1] | 83.9 [79.9 to 87.4] | 76.1 [71.5 to 80.3]
  B/Victoria (Day 22) | 99.9 [98.6 to 100] | 100 [99.1 to 100] | 99.5 [98.2 to 99.9] | 97.9 [95.9 to 99.1]
  B/Victoria (Day 181) | 95.3 [92.7 to 97.1] | 93.9 [91.1 to 96.1] | 86.7 [83.0 to 89.9] | 76.9 [72.2 to 80.9]

8. Secondary Outcome: Immunogenicity Endpoints: Percentage of Subjects With HI Titer ≥1:110, ≥1:151, ≥1:215, ≥1:330 and ≥1:629 on Day 22 Against Homologous Strains
Description: The percentage of subjects achieving HI Titers ≥1:110, ≥1:151, ≥1:215, ≥1:330 and ≥1:629 at Day 22 after vaccination is reported against homologous strains.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 22
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 398 | 397 | 389
percentage of subjects
  A/H1N1, HI ≥1:110 | 100.0 [99.1 to 100.0] | 100.0 [99.1 to 100.0] | 99.7 [98.6 to 100.0] | 97.7 [95.6 to 98.9]
  A/H1N1, HI ≥1:151 | 100.0 [99.1 to 100.0] | 100.0 [99.1 to 100.0] | 99.5 [98.2 to 99.9] | 97.4 [95.3 to 98.8]
  A/H1N1, HI ≥1:215 | 99.8 [98.6 to 100.0] | 99.2 [97.8 to 99.8] | 97.5 [95.4 to 98.8] | 93.8 [90.9 to 96.0]
  A/H1N1, HI ≥1:330 | 97.3 [95.2 to 98.6] | 93.7 [90.8 to 95.9] | 93.2 [90.3 to 95.5] | 82.5 [78.3 to 86.1]
  A/ H1N1 ≥1:629 | 94.8 [92.1 to 96.7] | 87.6 [84.0 to 90.7] | 87.9 [84.3 to 91.0] | 74.2 [69.6 to 78.5]
  A/H3N2, HI ≥1:110 | 99.8 [98.6 to 100.0] | 100.0 [99.1 to 100.0] | 100.0 [99.1 to 100.0] | 99.5 [98.1 to 99.9]
  A/H3N2, HI ≥1:151 | 99.8 [98.6 to 100.0] | 100.0 [99.1 to 100.0] | 100.0 [99.1 to 100.0] | 99.5 [98.1 to 99.9]
  A/H3N2, HI ≥1:215 | 99.5 [98.2 to 99.9] | 100.0 [99.1 to 100.0] | 100.0 [99.1 to 100.0] | 97.7 [95.6 to 98.9]
  A/H3N2, HI ≥1:330 | 99.3 [97.8 to 99.8] | 99.7 [98.6 to 100.0] | 99.5 [98.2 to 99.9] | 95.9 [93.4 to 97.6]
  A/H3N2, HI ≥1:629 | 99.0 [97.5 to 99.7] | 99.7 [98.6 to 100.0] | 99.2 [97.8 to 99.8] | 95.1 [92.4 to 97.0]
  B/Yamagata, HI ≥1:110 | 90.8 [87.5 to 93.4] | 88.4 [84.8 to 91.4] | 82.7 [78.6 to 86.3] | 68.3 [63.4 to 73.0]
  B/Yamagata, HI ≥1:151 | 87.6 [83.9 to 90.6] | 81.6 [77.4 to 85.3] | 75.9 [71.4 to 80.0] | 59.9 [54.8 to 64.9]
  B/Yamagata, HI ≥1:215 | 69.9 [65.2 to 74.3] | 64.2 [59.3 to 69.0] | 53.3 [48.2 to 58.3] | 38.5 [33.6 to 43.6]
  B/Yamagata, HI ≥1:330 | 44.0 [39.1 to 49.0] | 34.3 [29.6 to 39.2] | 25.1 [20.9 to 29.7] | 14.9 [11.5 to 18.9]
  B/Yamagata, HI ≥1:629 | 27.9 [23.5 to 32.5] | 20.9 [17.0 to 25.2] | 14.2 [10.9 to 18.1] | 7.3 [4.9 to 10.4]
  B/Victoria, HI ≥1:110 | 93.0 [90.1 to 95.3] | 89.9 [86.5 to 92.7] | 86.0 [82.8 to 89.8] | 76.1 [71.5 to 80.3]
  B/Victoria, HI ≥1:151 | 91.3 [88.1 to 93.9] | 87.9 [84.3 to 90.9] | 83.0 [78.9 to 86.6] | 70.6 [65.8 to 75.1]
  B/Victoria, HI ≥1:215 | 79.6 [75.3 to 83.4] | 73.4 [69.1 to 78.0] | 67.5 [62.6 to 72.1] | 53.0 [47.9 to 58.1]
  B/Victoria, HI ≥1:330 | 58.7 [53.7 to 63.6] | 48.7 [43.8 to 53.8] | 41.9 [37.0 to 46.9] | 32.0 [27.4 to 37.0]
  B/Victoria, HI ≥1:629 | 45.3 [40.3 to 50.3] | 37.6 [32.8 to 42.6] | 34.3 [29.6 to 39.2] | 24.1 [19.9 to 28.8]

9. Secondary Outcome: Immunogenicity Endpoint: GMT as Determined by HI Assay on Day 1, Day 22, and Day 181 Against Heterologous Strains
Description: GMT and 95% CI were analyzed for Day 22 for the heterologous strains using ANCOVA with study specific covariates.
  The two heterologous strains selected for HI testing in this study were the H3N2 strain, A/Hong Kong/4801/2014 (X-263B), and the B/ Victoria lineage strain, B/Malaysia/2506/2004.
Time Frame: Day 1, Day 22, Day 181
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 60 | 57 | 59 | 58
titer
  A/H3N2 (Day 1) | 97.7 [59.4 to 160.6] | 156.6 [96.1 to 255.1] | 40.9 [25.3 to 66.0] | 91.6 [55.6 to 150.8]
  A/H3N2 (Day 22) | 2436.1 [2058.0 to 2883.6] | 2415.2 [2049.9 to 2845.5] | 2225.1 [1872.6 to 2643.8] | 2097.2 [1769.7 to 2485.2]
  A/H3N2 (Day 181) | 898.1 [707.5 to 1139.9] | 917.6 [728.2 to 1156.3] | 953.2 [746.7 to 1216.6] | 791.7 [621.5 to 1008.3]
  B/Victoria (Day 1) | 33.4 [24.6 to 45.3] | 23.8 [17.6 to 32.2] | 15.8 [11.8 to 21.2] | 15.9 [11.7 to 21.6]
  B/Victoria (Day 22) | 327.1 [255.7 to 418.4] | 248.4 [195.3 to 316.0] | 283.2 [222.8 to 359.8] | 204.8 [159.6 to 262.8]
  B/Victoria (Day 181) | 107.1 [79.3 to 144.6] | 85.6 [63.9 to 114.7] | 77.5 [57.9 to 103.9] | 56.0 [41.2 to 76.0]

10. Secondary Outcome: Immunogenicity Endpoint: GMR as Determined by HI Assay for Day 22/Day 1 and Day 181/Day 1 Against Heterologous Strains
Description: The GMR is the geometric mean of the fold increase in HI titer from Day 1 to Day 22 or Day 181. GMR and 95% CI were analyzed for the heterologous strains using ANCOVA with study specific covariates.
  The two heterologous strains selected for HI testing in this study were the H3N2 strain, A/Hong Kong/4801/2014 (X-263B), and the B Victoria lineage strain, B/Malaysia/2506/2004.
Time Frame: Day 22/Day 1 and Day 181/Day 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 60 | 57 | 59 | 58
ratio
  A/H3N2 (Day 22/Day 1) | 14.67 [12.4 to 17.4] | 14.55 [12.3 to 17.1] | 13.40 [11.3 to 15.9] | 12.63 [10.7 to 15.0]
  A/H3N2 (Day 181/Day 1) | 5.31 [4.2 to 6.7] | 5.42 [4.3 to 6.8] | 5.63 [4.4 to 7.2] | 4.68 [3.7 to 6.0]
  B/Victoria (Day 22/Day 1) | 13.40 [10.5 to 17.1] | 10.18 [8.0 to 13.0] | 11.60 [9.1 to 14.7] | 8.39 [6.5 to 10.8]
  B/Victoria (Day 181/Day 1) | 4.38 [3.2 to 5.9] | 3.50 [2.6 to 4.7] | 3.17 [2.4 to 4.3] | 2.29 [1.7 to 3.1]

11. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving SCR and HI Titer ≥1:40 on Day 22 and Day 181 Against Heterologous Strains
Description: The percentage of subjects achieving HI titer ≥1:40 at Day 22 and Day 181 after vaccination and the percentage of subject who experienced seroconversion is reported for homologous strains. Seroconversion was defined in subjects seronegative at baseline (i.e. HI titer <1:10 on Day 1) as post-vaccination HI titer ≥1:40 and defined in subjects seropositive at baseline (i.e. HI titer ≥1:10 on Day 1) as a minimum of a 4-fold increase in post-vaccination HI titer.
  The two heterologous strains selected for HI testing in this study were the H3N2 strain, A/Hong Kong/4801/2014 (X-263B), and the B/Victoria lineage strain, B/Malaysia/2506/2004.
Time Frame: Day 22, Day 181
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 60 | 57 | 59 | 58
percentage of subjects
  A/H3N2, SCR (Day 22) | 78.3 [65.8 to 87.9] | 73.7 [60.3 to 84.5] | 83.1 [71.0 to 91.6] | 69.0 [55.5 to 80.5]
  A/ H3N2, HI titer ≥1:40 (Day 22) | 100 [94.0 to 100] | 100 [93.7 to 100] | 100 [93.9 to 100] | 100 [93.8 to 100]
  A/ H3N2, HI titer ≥1:40 (Day 181) | 100 [93.8 to 100] | 100 [93.68 to 100] | 100 [93.8 to 100] | 98.2 [90.4 to 100]
  B/Victoria, SCR (Day 22) | 75.0 [62.1 to 85.3] | 82.1 [69.6 to 91.1] | 81.4 [69.1 to 90.3] | 77.6 [64.7 to 87.5]
  B/Victoria, HI titer ≥1:40 (Day 22) | 98.3 [91.1 to 100] | 100 [93.6 to 100] | 96.6 [88.3 to 99.6] | 98.3 [90.8 to 100]
  B/ Victoria, HI titer ≥1:40 (Day 181) | 91.4 [81.0 to 97.1] | 83.6 [71.2 to 92.2] | 74.1 [61.0 to 84.7] | 64.3 [50.4 to 76.6]

12. Secondary Outcome: Immunogenicity Endpoint: GMT as Determined by Microneutralization (MN) Assay on Day 1, Day 22, and Day 181 Against Homologous Strains
Description: To further characterize immune response, MN GMT and 95% CI were analyzed for Day 1, Day 22, and Day 181 against homologous strains.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 1, Day 22, Day 181
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 60 | 60 | 60 | 60
titer
  A/H1N1 (Day 1) | 264.36 [173.8 to 402.1] | 198.13 [127.8 to 307.0] | 104.28 [67.0 to 162.3] | 140.38 [90.0 to 219.1]
  A/H1N1 (Day 22) | 2253.81 [1713.5 to 2964.5] | 2295.46 [1729.5 to 3046.7] | 2992.29 [2238.5 to 3999.9] | 1543.54 [1156.5 to 20660.1]
  A/H1N1 (Day 181) | 727.04 [568.6 to 929.6] | 725.35 [560.7 to 938.4] | 686.98 [527.2 to 895.2] | 412.34 [317.2 to 536.0]
  A/H3N2 (Day 1) | 160.88 [103.6 to 249.7] | 113.74 [71.9 to 180.0] | 133.25 [83.8 to 211.8] | 97.47 [61.1 to 155.6]
  A/H3N2 (Day 22) | 5532.06 [4441.7 to 6890.0] | 6649.94 [5275.3 to 8382.7] | 5019.51 [3978.6 to 6332.8] | 4696.37 [3699.4 to 5962.1]
  A/H3N2 (Day 181) | 2069.22 [1488.8 to 2875.9] | 2127.88 [1500.4 to 3017.8] | 2138.80 [1505.0 to 3039.5] | 1696.57 [1178.4 to 2442.5]
  B/Yamagata (Day 1) | 29.82 [22.2 to 40.1] | 37.99 [27.9 to 51.7] | 21.57 [15.8 to 29.5] | 21.07 [15.4 to 28.9]
  B/Yamagata (Day 22) | 388.29 [299.1 to 504.0] | 301.39 [229.0 to 396.7] | 247.31 [187.6 to 326.0] | 197.51 [149.3 to 261.4]
  B/Yamagata (Day 181) | 107.05 [81.4 to 140.8] | 103.59 [77.5 to 138.5] | 82.90 [61.9 to 111.0] | 56.03 [41.5 to 75.6]
  B/Victoria (Day 1) | 43.66 [33.1 to 57.6] | 43.13 [32.3 to 57.6] | 27.96 [20.9 to 37.4] | 33.14 [24.7 to 44.4]
  B/Victoria (Day 22) | 355.63 [271.8 to 465.4] | 346.99 [262.6 to 458.5] | 338.49 [255.0 to 449.4] | 193.09 [145.5 to 256.3]
  B/Victoria (Day 181) | 124.31 [95.3 to 162.1] | 106.08 [80.2 to 140.3] | 95.87 [72.1 to 127.5] | 60.54 [45.4 to 80.7]

13. Secondary Outcome: Immunogenicity Endpoint: GMR as Determined by MN Assay for Day 22/Day 1 and Day 181/Day 1 Against Homologous Strains
Description: The GMR is the geometric mean of the fold increase in MN titer from Day 1 to Day 22 or Day 181. GMR and 95% CI were analyzed for the homologous strains using ANCOVA with study specific covariates.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 22/Day 1 and Day 181/Day 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 60 | 60 | 60 | 60
ratio
  A/H1N1 (Day 22/Day 1) | 11.85 [9.0 to 15.6] | 12.07 [9.1 to 16.0] | 15.73 [11.8 to 21.0] | 8.11 [6.1 to 10.8]
  A/H1N1 (Day 181/Day 1) | 3.67 [2.9 to 4.7] | 3.66 [2.8 to 4.7] | 3.47 [2.7 to 4.5] | 2.08 [1.6 to 2.7]
  A/H3N2 (Day 22/Day 1) | 28.19 [22.6 to 35.1] | 33.88 [26.9 to 42.7] | 25.57 [20.3 to 32.3] | 23.93 [18.8 to 30.4]
  A/H3N2 (Day 181/Day 1) | 10.63 [7.6 to 14.8] | 10.93 [7.7 to 15.5] | 10.99 [7.7 to 15.6] | 8.72 [6.1 to 12.5]
  B/Yamagata (Day 22/Day 1) | 14.11 [10.9 to 18.3] | 10.95 [8.3 to 14.4] | 8.99 [6.8 to 11.8] | 7.18 [5.4 to 9.5]
  B/Yamagata (Day 181/Day 1) | 3.97 [3.0 to 5.2] | 3.84 [2.9 to 5.1] | 3.07 [2.3 to 4.1] | 2.08 [1.5 to 2.8]
  B/Victoria (Day 22/Day 1) | 9.43 [7.2 to 12.3] | 9.20 [7.0 to 12.2] | 8.97 [6.8 to 11.9] | 5.12 [3.9 to 6.8]
  B/Victoria (Day 181/Day 1) | 3.25 [2.5 to 4.2] | 2.77 [2.1 to 3.7] | 2.51 [1.9 to 3.3] | 1.58 [1.2 to 2.1]

14. Secondary Outcome: Immunogenicity Endpoint: Anti-neuraminidase (NA) GMTs on Day 1, Day 22, and Day 181 Against Homologous Strains
Description: To further characterize immune response, adjusted anti-NA GMT and 95% CI were analyzed for Day 1, Day 22, and Day 181 against homologous strains.
  Strains tested: N1 (PR8 H6N1 California/07/2009), N2 (PR8 H6N2 Switzerl/9715293/2013); B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 1, Day 22, Day 181
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 56 | 62 | 59 | 60
titer
  N1 (Day 1) | 1174.69 [767.8 to 1797.3] | 1209.21 [815.7 to 1792.6] | 230.09 [154.7 to 342.2] | 182.80 [122.7 to 272.2]
  N1 (Day 22) | 3403.72 [2821.4 to 4106.2] | 3161.01 [2654.7 to 3763.9] | 3588.43 [2994.0 to 4300.9] | 2410.65 [2001.2 to 2903.9]
  N1 (Day 181) | 2477.65 [1958.9 to 3133.7] | 1649.89 [1324.9 to 2054.5] | 2018.32 [1610.4 to 2529.5] | 870.73 [691.0 to 1097.2]
  N2 (Day 1) | 204.59 [121.3 to 345.2] | 289.86 [178.6 to 470.4] | 86.08 [52.8 to 140.3] | 86.34 [52.9 to 140.9]
  N2 (Day 22) | 915.19 [753.5 to 1111.6] | 1050.44 [876.7 to 1258.7] | 1242.36 [1031.4 to 1496.5] | 980.87 [813.8 to 1182.2]
  N2 (Day 181) | 505.91 [375.2 to 682.2] | 565.69 [426.7 to 749.9] | 516.51 [388.6 to 686.4] | 369.04 [277.5 to 490.8]
  B/Victoria (Day 1) | 497.11 [344.3 to 717.7] | 548.92 [390.7 to 771.2] | 306.48 [217.6 to 431.7] | 237.96 [168.7 to 335.6]
  B/Victoria (Day 22) | 3175.99 [2736.5 to 3686.0] | 3336.65 [2906.2 to 3830.8] | 3331.87 [2894.6 to 3835.2] | 2418.50 [2094.6 to 2792.74]
  B/Victoria (Day 181) | 1424.38 [1108.1 to 1831.0] | 1587.86 [1256.5 to 2006.6] | 1443.37 [1140.1 to 1827.3] | 1030.77 [810.3 to 1311.3]
  B/Yamagata (Day 1) | 290.06 [202.3 to 415.8] | 282.17 [201.7 to 394.8] | 148.35 [106.0 to 207.6] | 126.07 [90.0 to 176.6]
  B/Yamagata (Day 22) | 1288.67 [1094.6 to 1517.2] | 1250.88 [1074.3 to 1456.5] | 1275.06 [1093.5 to 1486.7] | 883.66 [756.1 to 1032.7]
  B/Yamagata (Day 181) | 727.17 [560.2 to 943.9] | 596.62 [467.2 to 762.0] | 511.73 [400.7 to 653.5] | 391.23 [305.3 to 501.3]

15. Secondary Outcome: Immunogenicity Endpoint: Anti-NA GMR for Day 22/Day 1 and Day 181/Day 1 Against Homologous Strains
Description: The GMR is the geometric mean of the fold increase in anti-NA titer from Day 1 to Day 22 or Day 181. GMR and 95% CI were analyzed against homologous strains using ANCOVA with study specific covariates.
  Strains tested: N1 (PR8 H6N1 California/07/2009), N2 (PR8 H6N2 Switzerl/9715293/2013); B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 22/Day 1 and Day 181/Day 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 56 | 62 | 59 | 60
ratio
  N1 (Day 22/Day 1) | 5.40 [4.5 to 6.5] | 5.02 [4.2 to 6.0] | 5.70 [4.8 to 6.8] | 3.83 [3.2 to 4.6]
  N1 (Day 181/Day 1) | 3.95 [3.1 to 5.0] | 2.63 [2.1 to 3.3] | 3.22 [2.6 to 4.0] | 1.39 [1.1 to 1.8]
  N2 (Day 22/Day 1) | 4.51 [3.7 to 5.5] | 5.18 [4.3 to 6.2] | 6.13 [5.1 to 7.4] | 4.84 [4.0 to 5.8]
  N2 (Day 181/Day 1) | 2.45 [1.8 to 3.3] | 2.74 [2.1 to 3.6] | 2.50 [1.9 to 3.3] | 1.79 [1.3 to 2.4]
  B/Yamagata (Day 22/Day 1) | 5.75 [4.9 to 6.8] | 5.59 [4.8 to 6.5] | 5.69 [4.9 to 6.6] | 3.95 [3.4 to 4.6]
  B/Yamagata (Day 181/Day 1) | 3.29 [2.5 to 4.3] | 2.70 [2.1 to 3.4] | 2.32 [1.81 to 3.0] | 1.77 [1.4 to 2.3]
  B/Victoria (Day 22/Day 1) | 6.81 [5.9 to 7.9] | 7.15 [6.2 to 8.2] | 7.14 [6.2 to 8.2] | 5.18 [4.5 to 6.0]
  B/Victoria (Day 181/Day 1) | 3.05 [2.4 to 3.9] | 3.40 [2.7 to 4.3] | 3.09 [2.4 to 3.9] | 2.21 [1.7 to 2.8]

16. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Solicited AEs
Description: Safety of revaccination was assessed in terms of percentage of subjects reporting solicited AEs up to 7 days after vaccination.
Time Frame: Day 1 to Day 7 after vaccination
Population: The solicited safety set consisting of all subjects who received a study vaccination with evaluable solicited AE data recorded on a diary card.
Measure: Number; unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 403 | 402 | 393
percentage of subjects
  Any Solicited AE | 64.76 | 50.12 | 53.48 | 40.71
  Solicited Local AE | 44.67 | 37.97 | 36.82 | 29.52
  Solicited Systemic AE | 39.21 | 24.81 | 30.85 | 18.83
  Other (analgesic/antipyretic use) | 27.54 | 10.17 | 16.92 | 10.43

17. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Unsolicited AEs
Description: Safety of revaccination was assessed in terms of percentage of subjects reporting unsolicited AEs during the overall study period (Day 1 to Day 366).
Time Frame: Day 1 to Day 366
Population: The unsolicited safety set consisting of all subjects who received a study vaccination with documented safety assessments for unsolicited AE data (including those where it was reported/confirmed that no events had occurred).
Measure: Number; unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 403 | 402 | 393
percentage of subjects
  Any Unsolicited AE | 54.09 | 55.33 | 55.97 | 52.16
  Related Unsolicited AE | 6.20 | 3.97 | 5.72 | 3.82

18. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Serious Adverse Events (SAE), AEs Leading to Withdrawal, New Onset of Chronic Disease (NOCD), AE of Special Interest (AESI), and Medically Attended AE.
Description: Safety of revaccination was assessed in terms of percentage of subjects reporting SAEs, AEs leading to withdrawal, NOCD, AESI and medically attended AE. Each subject was followed for a period of 12 months after receipt of the study vaccine.
  NOCDs include AEs that represents a new diagnosis of a chronic medical condition that was not present or suspected in a subject prior to study enrollment. AESIs include potentially immune-mediated disorders which were reported by the investigators.
Time Frame: Day 1 to Day 366
Population: The unsolicited safety set consisting of all subjects who received a study vaccination with documented safety assessments for unsolicited adverse event (AE) data (including those where it was reported/confirmed that no events had occurred).
Measure: Number; unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 403 | 402 | 393
percentage of subjects
  SAE | 2.48 | 2.73 | 1.74 | 2.04
  AE leading to withdrawal | 0 | 0 | 0 | 0
  NOCD | 0.50 | 0 | 0 | 0
  AESI | 0 | 0 | 0 | 0.25
  Medically attended AE | 51.61 | 54.34 | 53.98 | 48.60

19. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Diagnosis of Failure to Thrive or Short Stature
Description: Safety of revaccination was assessed in terms of percentage of subjects reporting diagnosis of failure to thrive or short stature up to 12 months after last vaccination.
Time Frame: Day 1 to Day 366
Population: as for outcome 17
Measure: Number; unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 403 | 402 | 393
percentage of subjects | 0.25 | 0.74 | 0.25 | 0.76

20. Secondary Outcome: Safety Endpoint: Percentage of Subjects With Otitis Media, or Pneumonia, or Influenza-like Illness
Description: Safety of revaccination was assessed in terms of percentage of subjects reporting otitis media, or pneumonia, or influenza-like illness up to 12 months after last vaccination.
Time Frame: Day 1 to Day 366
Population: as for outcome 17
Measure: Number; unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 403 | 403 | 402 | 393
percentage of subjects
  otitis media, any event | 3.23 | 3.47 | 3.73 | 2.80
  pneumonia, any event | 1.49 | 1.49 | 0.75 | 1.78
  influenza-like illness | 7.94 | 10.17 | 9.20 | 7.89

21. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects With MN Titer ≥1:20, ≥1:40, ≥1:80, ≥1:160, ≥1:320 and ≥1:640 on Day 22 and Day 181 Against Homologous Strains
Description: The percentage of subjects achieving MN titer ≥1:20, ≥1:40, ≥1:80 ≥1:160, ≥1:320 and ≥1:640 at Day 22 and Day 181 after vaccination is reported against homologous strains.
  Strains tested: A/H1N1 California/07/2009; A/H3N2 Switzerland/9715293/2013; B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 22, Day 181
Population: The Immunogenicity PPS consisting of all subjects who received a study vaccination and provided immunogenicity data (MN titer ≥1:20, ≥1:40, ≥1:80, >four-fold rise), and who correctly received the study vaccine, had no major protocol deviations, and did not develop RT-PCR-confirmed influenza infection between baseline and Visit 2.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 60 | 59 | 60 | 59
percentage of subjects
  A/ H1N1, ≥1:20 (Day 22) | 100.00 [93.94 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 100.00 [93.94 to 100.00]
  A/ H1N1, ≥1:40 (Day 22) | 98.31 [90.91 to 99.96] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 100.00 [93.94 to 100.00]
  A/H1N1, ≥1:80 (Day 22) | 98.31 [90.91 to 99.96] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 98.31 [90.91 to 99.96]
  A/H1N1, ≥1:160 (Day 22) | 98.31 [90.91 to 99.96] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 94.92 [85.85 to 98.94]
  A/H1N1, ≥1:320 (Day 22) | 96.61 [88.29 to 99.59] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 94.92 [85.85 to 98.94]
  A/H1N1, ≥1:640 (Day 22) | 96.61 [88.29 to 99.59] | 98.31 [90.91 to 99.96] | 91.67 [81.61 to 97.24] | 81.36 [69.09 to 90.31]
  A/H1N1, ≥1:20 (Day 181) | 100.00 [94.04 to 100.00] | 100.00 [93.84 to 100.00] | 100.00 [93.84 to 100.00] | 98.28 [90.76 to 99.96]
  A/H1N1, ≥1:40 (Day 181) | 100.00 [94.04 to 100.00] | 100.00 [93.84 to 100.00] | 100.00 [93.84 to 100.00] | 96.55 [88.09 to 99.58]
  A/H1N1, ≥1:80 (Day 181) | 100.00 [94.04 to 100.00] | 100.00 [93.84 to 100.00] | 100.00 [93.84 to 100.00] | 93.10 [83.27 to 98.09]
  A/H1N1, ≥1:160 (Day 181) | 96.67 [88.47 to 99.59] | 98.28 [90.76 to 99.96] | 94.83 [85.62 to 98.92] | 81.03 [68.59 to 90.13]
  A/H1N1, ≥1:320 (Day 181) | 91.67 [81.61 to 97.24] | 91.38 [81.02 to 97.14] | 84.48 [72.58 to 92.65] | 63.79 [50.12 to 76.01]
  A/H1N1, ≥1:640 (Day 181) | 80.00 [67.67 to 89.22] | 63.79 [50.12 to 76.01] | 55.17 [41.54 to 68.26] | 48.28 [34.95 to 61.78]
  A/H3N2, ≥1:20 (Day 22) | 100.00 [94.04 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 98.28 [90.76 to 99.96]
  A/H3N2, ≥1:40 (Day 22) | 100.00 [94.04 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 98.28 [90.76 to 99.96]
  A/H3N2, ≥1:80 (Day 22) | 100.00 [94.04 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 98.28 [90.76 to 99.96]
  A/H3N2, ≥1:160 (Day 22) | 100.00 [94.04 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 98.28 [90.76 to 99.96]
  A/H3N2, ≥1:320 (Day 22) | 100.00 [94.04 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 98.28 [90.76 to 99.96]
  A/H3N2, ≥1:640 (Day 22) | 100.00 [94.04 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 98.28 [90.76 to 99.96]
  A/H3N2, ≥1:20 (Day 181) | 100.00 [94.04 to 100.00] | 98.28 [90.76 to 99.96] | 100.00 [93.84 to 100.00] | 98.21 [90.45 to 99.95]
  A/H3N2, ≥1:40 (Day 181) | 100.00 [94.04 to 100.00] | 98.28 [90.76 to 99.96] | 100.00 [93.84 to 100.00] | 96.43 [87.69 to 99.56]
  A/H3N2, ≥1:80 (Day 181) | 100.00 [94.04 to 100.00] | 98.28 [90.76 to 99.96] | 100.00 [93.84 to 100.00] | 91.07 [80.38 to 97.04]
  A/H3N2, ≥1:160 (Day 181) | 96.67 [88.47 to 99.59] | 98.28 [90.76 to 99.96] | 96.55 [88.09 to 99.58] | 89.29 [78.12 to 95.97]
  A/H3N2, ≥1:320 (Day 181) | 91.67 [81.61 to 97.24] | 94.83 [85.62 to 98.92] | 93.10 [83.27 to 98.09] | 85.71 [73.78 to 93.62]
  A/H3N2, ≥1:640 (Day 181) | 86.67 [75.41 to 94.06] | 86.21 [74.62 to 93.85] | 84.48 [72.58 to 92.65] | 83.93 [71.67 to 92.38]
  B/Yamagata, ≥1:20 (Day 22) | 100.00 [94.04 to 100.00] | 100.00 [93.94 to 100.00] | 96.67 [88.47 to 99.59] | 96.55 [88.09 to 99.58]
  B/Yamagata, ≥1:40 (Day 22) | 98.33 [91.06 to 99.96] | 98.31 [90.91 to 99.96] | 96.67 [88.47 to 99.59] | 93.10 [83.27 to 98.09]
  B/Yamagata, ≥1:80 (Day 22) | 95.00 [86.08 to 98.96] | 96.61 [88.29 to 99.59] | 95.00 [86.08 to 98.96] | 89.66 [78.83 to 96.11]
  B/Yamagata, ≥1:160 (Day 22) | 91.67 [81.61 to 97.24] | 86.44 [75.02 to 93.96] | 78.33 [65.80 to 87.93] | 70.69 [57.27 to 81.91]
  B/Yamagata, ≥1:320 (Day 22) | 75.00 [62.14 to 85.28] | 72.88 [59.73 to 83.64] | 65.00 [51.60 to 76.87] | 50.00 [36.58 to 63.42]
  B/Yamagata, ≥1:640 (Day 22) | 58.33 [44.88 to 70.93] | 47.46 [34.30 to 60.88] | 31.67 [20.26 to 44.96] | 24.14 [13.87 to 37.17]
  B/Yamagata, ≥1:20 (Day 181) | 98.33 [91.06 to 99.96] | 96.55 [88.09 to 99.58] | 93.10 [83.27 to 98.09] | 80.36 [67.57 to 89.77]
  B/Yamagata, ≥1:40 (Day 181) | 93.33 [83.80 to 98.15] | 93.10 [83.27 to 98.09] | 79.31 [66.65 to 88.83] | 71.43 [57.79 to 82.70]
  B/Yamagata, ≥1:80 (Day 181) | 71.67 [58.56 to 82.55] | 72.41 [59.10 to 83.34] | 56.90 [42.23 to 69.84] | 46.43 [32.99 to 60.26]
  B/Yamagata, ≥1:160 (Day 181) | 45.00 [32.12 to 58.39] | 48.28 [34.95 to 61.78] | 32.76 [21.01 to 46.34] | 17.86 [8.91 to 30.40]
  B/Yamagata, ≥1:320 (Day 181) | 25.00 [14.72 to 37.86] | 24.14 [13.87 to 37.17] | 15.52 [7.35 to 27.42] | 7.14 [1.98 to 17.29]
  B/Yamagata, ≥1:640 (Day 181) | 3.33 [0.41 to 11.53] | 8.62 [2.86 to 18.98] | 5.17 [1.08 to 14.38] | 3.57 [0.44 to 12.31]
  B/Victoria, ≥1:20 (Day 22) | 98.31 [90.91 to 99.96] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00] | 98.31 [90.91 to 99.96]
  B/Victoria, ≥1:40 (Day 22) | 94.92 [85.85 to 98.94] | 100.00 [93.94 to 100.00] | 96.67 [88.47 to 99.59] | 93.22 [83.54 to 98.12]
  B/Victoria, ≥1:80 (Day 22) | 91.53 [81.32 to 97.19] | 96.61 [88.29 to 99.59] | 90.00 [79.49 to 96.24] | 84.75 [73.01 to 92.78]
  B/Victoria, ≥1:160 (Day 22) | 86.44 [75.02 to 93.96] | 86.44 [75.02 to 93.96] | 81.67 [69.56 to 90.48] | 69.49 [56.13 to 80.81]
  B/Victoria, ≥1:320 (Day 22) | 74.58 [61.56 to 85.02] | 67.80 [54.36 to 79.38] | 58.33 [44.88 to 70.93] | 35.59 [23.55 to 49.13]
  B/Victoria, ≥1:640 (Day 22) | 49.15 [35.89 to 62.50] | 42.37 [29.61 to 55.93] | 33.33 [21.69 to 46.69] | 22.03 [12.29 to 34.73]
  B/Victoria, ≥1:20 (Day 181) | 100.00 [94.04 to 100.00] | 100.00 [93.84 to 100.00] | 98.28 [90.76 to 99.96] | 96.43 [87.69 to 99.56]
  B/Victoria, ≥1:40 (Day 181) | 86.67 [75.41 to 94.06] | 87.93 [76.70 to 95.01] | 74.14 [60.96 to 84.74] | 60.71 [46.75 to 73.50]
  B/Victoria, ≥1:80 (Day 181) | 78.33 [65.80 to 87.93] | 63.79 [50.12 to 76.01] | 44.83 [31.74 to 58.46] | 41.07 [28.10 to 55.02]
  B/Victoria, ≥1:160 (Day 181) | 58.33 [44.88 to 70.93] | 43.10 [30.16 to 56.77] | 27.59 [16.66 to 40.90] | 23.21 [12.98 to 36.42]
  B/Victoria, ≥1:320 (Day 181) | 31.67 [20.26 to 44.96] | 20.69 [11.17 to 33.35] | 18.97 [9.87 to 31.41] | 8.93 [2.96 to 19.62]
  B/Victoria, ≥1:640 (Day 181) | 8.33 [2.76 to 18.39] | 15.52 [7.35 to 27.42] | 12.07 [4.99 to 23.30] | 5.36 [1.12 to 14.87]

22. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving Anti-NA Titers ≥1:20, ≥1:40, ≥1:80, ≥1:160, ≥1:320 and ≥1:640 on Days 22 and 181 Against Homologous Strains
Description: The percentage of subjects achieving anti-NA titers ≥1:20, ≥1:40, ≥1:80, ≥1:160, ≥1:320 and ≥1:640 on Days 22 and 181 after vaccination is reported against homologous strains
  Strains tested: N1 (PR8 H6N1 California/07/2009), N2 (PR8 H6N2 Switzerl/9715293/2013); B/Victoria Brisbane/60/2008; B/Yamagata Phuket/3073/2013.
Time Frame: Day 22, Day 181
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV/aQIV | aQIV/QIV | QIV/aQIV | QIV/QIV
Number analyzed (Participants) | 56 | 62 | 59 | 60
percentage of subjects
  N1, ≥1:20 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00]
  N1, ≥1:40 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 98.33 [91.06 to 99.96]
  N1, ≥1:80 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 98.33 [91.06 to 99.96]
  N1, ≥1:160 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 93.33 [83.80 to 98.15]
  N1, ≥1:320 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 88.33 [77.43 to 95.18]
  N1,≥1:640 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 98.31 [90.91 to 99.96] | 85.00 [73.43 to 92.90]
  N1, ≥1:20 (Day 181) | 100.00 [93.51 to 100.00] | 100.00 [94.13 to 100.00] | 100.00 [93.84 to 100.00] | 93.33 [83.80 to 98.15]
  N1, ≥1:40 (Day 181) | 100.00 [93.51 to 100.00] | 100.00 [94.13 to 100.00] | 100.00 [93.84 to 100.00] | 91.67 [81.61 to 97.24]
  N1, ≥1:80 (Day 181) | 100.00 [93.51 to 100.00] | 100.00 [94.13 to 100.00] | 100.00 [93.84 to 100.00] | 86.67 [75.41 to 94.06]
  N1, ≥1:160 (Day 181) | 100.00 [93.51 to 100.00] | 100.00 [94.13 to 100.00] | 96.55 [88.09 to 99.58] | 81.67 [69.56 to 90.48]
  N1, ≥1:320 (Day 181) | 100.00 [93.51 to 100.00] | 96.72 [88.65 to 99.60] | 93.10 [83.27 to 98.09] | 70.00 [56.79 to 81.15]
  N1, ≥1:640 (Day 181) | 100.00 [93.51 to 100.00] | 93.44 [84.05 to 98.18] | 72.41 [59.10 to 83.34] | 51.67 [38.39 to 64.77]
  N2, ≥1:20 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00]
  N2, ≥1:40 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00]
  N2, ≥1:80 (Day 22) | 98.21 [90.45 to 99.95] | 100.00 [94.22 to 100.00] | 98.31 [90.91 to 99.96] | 96.67 [88.47 to 99.59]
  N2, ≥1:160 (Day 22) | 98.21 [90.45 to 99.95] | 100.00 [94.22 to 100.00] | 98.31 [90.91 to 99.96] | 90.00 [79.49 to 96.24]
  N2, ≥1:320 (Day 22) | 94.64 [85.13 to 98.88] | 96.77 [88.83 to 99.61] | 94.92 [85.85 to 98.94] | 85.00 [73.43 to 92.90]
  N2, ≥1:640 (Day 22) | 85.71 [73.78 to 93.62] | 88.71 [78.11 to 95.34] | 79.66 [67.17 to 89.02] | 68.33 [55.04 to 79.74]
  N2, ≥1:20 (Day 181) | 100.00 [93.51 to 100.00] | 100.00 [94.04 to 100.00] | 100.00 [93.84 to 100.00] | 90.00 [79.49 to 96.24]
  N2, ≥1:40 (Day 181) | 98.18 [90.28 to 99.95] | 98.33 [91.06 to 99.96] | 89.66 [78.83 to 96.11] | 88.33 [77.43 to 95.18]
  N2, ≥1:80 (Day 181) | 94.55 [84.88 to 98.86] | 98.33 [91.06 to 99.96] | 86.21 [74.62 to 93.85] | 80.00 [67.67 to 89.22]
  N2, ≥1:160 (Day 181) | 85.45 [73.34 to 93.50] | 95.00 [86.08 to 98.96] | 81.03 [68.59 to 90.13] | 70.00 [56.79 to 81.15]
  N2, ≥1:320 (Day 181) | 80.00 [67.03 to 89.57] | 85.00 [73.43 to 92.90] | 67.24 [53.66 to 78.99] | 61.67 [48.21 to 73.93]
  N2, ≥1:640 (Day 181) | 70.91 [57.10 to 82.37] | 81.67 [69.56 to 90.48] | 55.17 [41.54 to 68.26] | 50.00 [36.81 to 63.19]
  B/Yamagata, ≥1:20 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.13 to 100.00] | 100.00 [93.04 to 100.00] | 100.00 [94.04 to 100.00]
  B/Yamagata, ≥1:40 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.13 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00]
  B/Yamagata, ≥1:80 (Day 22) | 98.21 [90.45 to 99.95] | 100.00 [94.13 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00]
  B/Yamagata, ≥1:160 (Day 22) | 98.21 [90.45 to 99.95] | 100.00 [94.13 to 100.00] | 100.00 [93.94 to 100.00] | 98.33 [91.06 to 99.96]
  B/Yamagata, ≥1:320 (Day 22) | 98.21 [90.45 to 99.95] | 100.00 [94.13 to 100.00] | 96.61 [88.29 to 99.59] | 88.33 [77.43 to 95.18]
  B/Yamagata, ≥1:640 (Day 22) | 91.07 [80.38 to 97.04] | 91.80 [81.90 to 97.28] | 89.83 [79.17 to 96.18] | 66.67 [53.31 to 78.31]
  B/Yamagata, ≥1:20 (Day 181) | 100.00 [93.51 to 100.00] | 98.33 [91.06 to 99.96] | 100.00 [93.84 to 100.00] | 100.00 [94.04 to 100.00]
  B/Yamagata, ≥1:40 (Day 181) | 100.00 [93.51 to 100.00] | 98.33 [91.06 to 99.96] | 98.28 [90.76 to 99.96] | 96.67 [88.47 to 99.59]
  B/Yamagata, ≥1:80 (Day 181) | 100.00 [93.51 to 100.00] | 98.33 [91.06 to 99.96] | 96.55 [88.09 to 99.58] | 90.00 [79.49 to 96.24]
  B/Yamagata, ≥1:160 (Day 181) | 98.18 [90.28 to 99.95] | 96.67 [88.47 to 99.59] | 91.38 [81.02 to 97.14] | 81.67 [69.56 to 90.48]
  B/Yamagata, ≥1:320 (Day 181) | 92.73 [82.41 to 97.98] | 86.67 [75.41 to 94.06] | 84.48 [72.58 to 92.65] | 65.00 [51.60 to 76.87]
  B/Yamagata, ≥1:640 (Day 181) | 72.73 [59.04 to 83.86] | 61.67 [48.21 to 73.93] | 51.72 [38.22 to 65.05] | 40.00 [27.56 to 53.46]
  B/Victoria, ≥1:20 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00]
  B/Victoria, ≥1:40 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00]
  B/Victoria, ≥1:80 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00]
  B/Victoria, ≥1:160 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 100.00 [94.04 to 100.00]
  B/Victoria, ≥1:320 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 98.33 [91.06 to 99.96]
  B/Victoria, ≥1:640 (Day 22) | 100.00 [93.62 to 100.00] | 100.00 [94.22 to 100.00] | 100.00 [93.94 to 100.00] | 91.67 [81.61 to 97.24]
  B/Victoria, ≥1:20 (Day 181) | 100.00 [93.51 to 100.00] | 100.00 [94.13 to 100.00] | 100.00 [93.84 to 100.00] | 100.00 [94.04 to 100.00]
  B/Victoria, ≥1:40 (Day 181) | 100.00 [93.51 to 100.00] | 100.00 [94.13 to 100.00] | 100.00 [93.84 to 100.00] | 100.00 [94.04 to 100.00]
  B/Victoria, ≥1:80 (Day 181) | 100.00 [93.51 to 100.00] | 100.00 [94.13 to 100.00] | 100.00 [93.84 to 100.00] | 100.00 [94.04 to 100.00]
  B/Victoria, ≥1:160 (Day 181) | 100.00 [93.51 to 100.00] | 100.00 [94.13 to 100.00] | 96.55 [88.09 to 99.58] | 96.67 [88.47 to 99.59]
  B/Victoria, ≥1:320 (Day 181) | 94.55 [84.88 to 98.86] | 100.00 [94.13 to 100.00] | 95.55 [88.09 to 99.58] | 83.33 [71.48 to 91.71]
  B/Victoria, ≥1:640 (Day 181) | 89.09 [77.75 to 95.89] | 95.08 [86.29 to 98.97] | 81.03 [68.59 to 90.13] | 70.00 [56.79 to 81.15]

ADVERSE EVENTS:
Time Frame: Day 1 - Day 366
Description: The overall safety set included all subjects who were in the solicited safety set and/or in the unsolicited safety set.
  Assessment of revaccination safety included:
  SAEs collected between Day 1 to Day 366 Non-serious AEs included solicited AEs collected between Day 1 to Day 7 after last vaccination, and unsolicited AEs collected between Day 1 to Day 366 after last vaccination
Groups:
- aQIV-aQIV: Subjects previously vaccinated with aQIV followed one year later by aQIV
  Adjuvanted QIV (aQIV): Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine (aQIV)
- aQIV-QIV: Subjects previously vaccinated with aQIV followed one year later by QIV
  Non-adjuvanted QIV: Non-adjuvanted Quadrivalent Influenza Vaccine (QIV)
- QIV-aQIV: Subjects previously vaccinated with QIV followed one year later by aQIV
  Adjuvanted QIV (aQIV): Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine (aQIV)
- QIV-QIV: Subjects previously vaccinated with QIV followed one year later by QIV
  Non-adjuvanted QIV: Non-adjuvanted Quadrivalent Influenza Vaccine (QIV)
Arm/Group | aQIV-aQIV | aQIV-QIV | QIV-aQIV | QIV-QIV
All-Cause Mortality (participants affected / at risk) | 0/403 | 0/403 | 0/402 | 0/393
Serious Adverse Events (participants affected / at risk) | 10/403 | 11/403 | 7/402 | 8/393
Other Adverse Events (participants affected / at risk) | 289/403 | 269/403 | 274/402 | 229/393
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV-aQIV (N=403) | aQIV-QIV (N=403) | QIV-aQIV (N=402) | QIV-QIV (N=393)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Spina Bifida Occulta (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 1
Amoebic Dysentery (Infections and infestations) | 1 | 0 | 0 | 0
Appendiceal Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Dengue Fever (Infections and infestations) | 1 | 0 | 0 | 0
External Ear Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 4 | 4 | 1
Herpangina (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1
Animal Bite (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Jaw Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound Secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Febrile Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Kawasaki's Disease (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV-aQIV (N=403) | aQIV-QIV (N=403) | QIV-aQIV (N=402) | QIV-QIV (N=393)
Diarrhoea (Gastrointestinal disorders) | 22 | 8 | 14 | 16
Vomiting (Gastrointestinal disorders) | 29 | 15 | 19 | 13
Influenza Like Illness (General disorders) | 32 | 41 | 37 | 31
Injection Site Erythema (General disorders) | 81 | 57 | 51 | 39
Injection Site Induration (General disorders) | 62 | 55 | 38 | 24
Injection Site Pain (General disorders) | 163 | 137 | 134 | 120
Pyrexia (General disorders) | 96 | 46 | 72 | 51
Nasopharyngitis (Infections and infestations) | 21 | 19 | 26 | 16
Upper Respiratory Tract Infection (Infections and infestations) | 78 | 100 | 99 | 73
Somnolence (Nervous system disorders) | 79 | 45 | 55 | 25
Eating Disorder (Psychiatric disorders) | 66 | 28 | 52 | 24
Irritability (Psychiatric disorders) | 60 | 44 | 50 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less